CLINICAL TRIAL: NCT03590756
Title: Influence of Mango Intake on Skin Health in Postmenopausal Women
Brief Title: Influence of Mango Intake of Skin Health in Postmenopausal Women
Acronym: MSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1185928
Record Dates: First submitted 2018-07-03; First posted 2018-07-18 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Wrinkle; Skin Red
Keywords: Skin Health; Skin Wrinkle; Skin Redness; Carotenoid; Mango
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High mango group (Experimental): 250g (1.5 cup) of mango intake per day, 4 days a week for 16 weeks
  Interventions: Other: 16 weeks mango intake
- Low mango group (Other): 85g (0.5 cup) of mango intake per day, 4 days a week for 16 weeks
  Interventions: Other: 16 weeks mango intake

INTERVENTIONS:
Other: 16 weeks mango intake — Participants will be provided fresh frozen Ataulfo mangoes.

SUMMARY:
This study aims to investigate the effects on 16 weeks of mango intake on skin health in postmenopausal women. Half of the participants will receive 85g portions of mangoes while the other half receive 250g portions of mangos. Participants will be instructed to consume the specific portion 4 times a week, for a total duration of 16 weeks.

DETAILED DESCRIPTION:
Mangoes are rich in carotenoids, flavonoids, vitamins and other active phytochemicals such as resistant starches. Although a role of mangoes in skin health has long been advocated in traditional medicine, little scientific research has been conducted.

We hypothesize that 85g (0.5 cups) of mango intake for 16 weeks will have minimal impact on skin health, while 250g (1.5 cups) of mango intake will produce significant benefits.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Fitzpatrick skin type I and II
* BMI 18.5 - 35.0 kg/m2
* Normal blood levels in the comprehensive metabolic panel, or values slightly out of range as approved by the study physician

Exclusion Criteria:

* Allergic to mangoes
* Fruit consumption of 2 or more cups per day
* Vegetable consumption of 3 or more cups per day for females
* Fruit juice consumption of more than 1 cup per day
* Self-reported malabsorption
* Currently taking regular prescription drugs i.e. statins, thyroid, anti-inflammatory drugs
* Had any medical or cosmetic procedures such as laser resurfacing or plastic surgery to the face within the last 6 months, including botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
* Autoimmune photosensitive condition or known genetic condition with a deficiency in collagen production (such as Ehler-Danlos)
* Smoking (current smoker, smoked within the past year, former smokers with greater than a 20 pack-year history of smoking within the past 20 years.
* Indications of substance or alcohol abuse
* Unwillingness to discontinue high antioxidant supplements during washout and interventions

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Skin Wrinkle Depth and Redness | 0, 8, and 16 week
  Using a skin camera from BrighTex Bio-Photonics to measure change in skin wrinkle depth and redness within a period of 16 weeks.
Skin carotenoid | 0, 4, 8, 12, and 16 weeks
  Using a skin photometer (Veggie Meter) to measure change in skin carotenoid within a period of 16 weeks.

SECONDARY OUTCOMES:
Sebum | 0, 8, 16, weeks
  Sebum will be collected with sebutapes from the face and stored for possible further analysis.
Plasma carotenoid | 0, 8, 16 weeks.
  Plasma samples will be collected and stored at -80C for possible further analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No